CLINICAL TRIAL: NCT02657837
Title: Measures of Respiratory Health
Brief Title: Measures of Respiratory Health (MRH)
Acronym: MRH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Other Study IDs: 1000051399
Record Dates: First submitted 2016-01-08; First posted 2016-01-18 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis; Asthma; Sickle Cell Anemia; Bronchiolitis Obliterans
Keywords: CF; Multiple Breath Washout; Lung Clearance Index; Pediatrics
MeSH Terms: conditions — Cystic Fibrosis; Asthma; Anemia, Sickle Cell; Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cystic Fibrosis: Children 2.5 to 18 years old with confirmed diagnosis of cystic fibrosis
- Children with other respiratory disease: Children 2.5 to 18 years old with confirmed diagnosis of respiratory disease including but not limited to asthma, transplant, and sickle cell anemia.
- Healthy Children: Children and adults 2.5 to 30 years old with no history of chronic disease

SUMMARY:
The Lung Clearance Index, measured by multiple breath washout, is a measure of lung function that is considered a research tool in Canada as the device used to measure it is not approved by Health Canada. The study will assess lung function in patients undergoing routine lung function testing for clinical indications (Cystic Fibrosis and Other Respiratory Diseases). In addition, healthy controls of different ages will be asked to perform this lung function test to gain reference data that can be used to interpret LCI in patients with lung disease.

DETAILED DESCRIPTION:
Functional abnormalities associated with lung disease such as cystic fibrosis (CF) occur in early childhood, but have historically gone undetected until the onset of clinical symptoms, at which point irreversible lung damage may have already occurred (1-3). Consequently, over the last ten years the focus of clinical care has shifted to early intervention and prevention of these structural changes. To facilitate early intervention there is a pressing need for surrogate markers of early obstructive lung disease that are also sensitive enough to detect treatment effects (4).

The Lung Clearance Index (LCI) is a promising marker for detecting early lung disease. The LCI is measured by multiple breath washout (MBW) and is an indicator of ventilation inhomogeneity. MBW is performed during quiet tidal breathing and requires minimal effort from patients. It is feasible in all age groups when adaptions are made for younger children.

While there are Health Canada licensed washout systems available that can determine LCI; these devices have not been adequately validated; thus their use in routine lung function testing is controversial. As part of an international effort to validate multiple breath washout testing to measure LCI, the specific device is licensed in Europe, but as of yet is not Health Canada approved. Thus, testing with this device is considered research. This study will utilize technology to assess lung function in patients undergoing routine lung function testing for clinical indications. In addition, healthy controls of different ages will be asked to perform this lung function test to gain reference data that can be used to interpret LCI in patients with lung disease.

ELIGIBILITY:
Participants with CF

Inclusion criteria:

1. 2.5 - 18 years of age at enrolment
2. Diagnosis of CF as evidenced by one or more clinical feature consistent with the CF phenotype or positive CF newborn screen AND one or more of the following criteria:

   1. A documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis (QPIT)
   2. A documented genotype with two disease-causing mutations in the CFTR gene
3. Informed consent by participant, parent, or legal guardian
4. Ability to perform technically acceptable MBW measurements

Exclusion criteria:

1. Physical findings at screening that would compromise the safety of the participant as judged by the patient's most responsible physician
2. Requirement of supplementary oxygen to maintain an oxygen saturation above 95%

Participants with other respiratory disease

Inclusion criteria:

1. MD diagnosed lung disease and/or attending the Pulmonary Function Laboratory
2. 2.5 - 18 years of age at enrollment
3. Informed consent by participant, parent, or legal guardian
4. Ability to perform technically acceptable MBW measurements

Exclusion criteria:

1. Physical findings at screening that would compromise the safety of the participant or the quality of the study data.
2. Requirement of supplementary oxygen to maintain an oxygen saturation above 95%

Healthy Participants

Inclusion criteria:

1. 2.5 - 30 years of age at enrollment
2. Informed consent by participant, parent, or legal guardian
3. Ability to perform technically acceptable MBW measurements

Exclusion criteria:

1. Physical findings at screening that would compromise the safety of the participant or the quality of the study data.
2. Evidence of a chronic disease process such as lung disease

Ages: 30 Months to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants who meet all of the inclusion and none of the exclusion criteria will be eligible for participation in this study. Participants will include individuals with CF, individuals with other respiratory disease and healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01; Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an abnormal Lung Clearance Index (>7.5). | Day 1
  Single time point measurements obtained in enrolled subjects

SECONDARY OUTCOMES:
. Proportion of patients with an abnormal pulmonary function tests based on spirometry. | Day 1
  Single time point measurements obtained in enrolled subjects

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Grasemann H, Ratjen F. Early lung disease in cystic fibrosis. Lancet Respir Med. 2013 Apr;1(2):148-57. doi: 10.1016/S2213-2600(13)70026-2. Epub 2013 Mar 12. PMID 24429095
- [Background] Ranganathan SC, Dezateux C, Bush A, Carr SB, Castle RA, Madge S, Price J, Stroobant J, Wade A, Wallis C, Stocks J; London Collaborative Cystic Fibrosis Group. Airway function in infants newly diagnosed with cystic fibrosis. Lancet. 2001 Dec 8;358(9297):1964-5. doi: 10.1016/s0140-6736(01)06970-7. PMID 11747924
- [Background] Sly PD, Brennan S, Gangell C, de Klerk N, Murray C, Mott L, Stick SM, Robinson PJ, Robertson CF, Ranganathan SC; Australian Respiratory Early Surveillance Team for Cystic Fibrosis (AREST-CF). Lung disease at diagnosis in infants with cystic fibrosis detected by newborn screening. Am J Respir Crit Care Med. 2009 Jul 15;180(2):146-52. doi: 10.1164/rccm.200901-0069OC. Epub 2009 Apr 16. PMID 19372250
- [Background] Horsley A. Lung clearance index in the assessment of airways disease. Respir Med. 2009 Jun;103(6):793-9. doi: 10.1016/j.rmed.2009.01.025. Epub 2009 Feb 25. PMID 19246184
- [Background] Gustafsson PM, Aurora P, Lindblad A. Evaluation of ventilation maldistribution as an early indicator of lung disease in children with cystic fibrosis. Eur Respir J. 2003 Dec;22(6):972-9. doi: 10.1183/09031936.03.00049502. PMID 14680088
- [Background] Aurora P, Gustafsson P, Bush A, Lindblad A, Oliver C, Wallis CE, Stocks J. Multiple breath inert gas washout as a measure of ventilation distribution in children with cystic fibrosis. Thorax. 2004 Dec;59(12):1068-73. doi: 10.1136/thx.2004.022590. PMID 15563707
- [Background] Gustafsson PM, De Jong PA, Tiddens HA, Lindblad A. Multiple-breath inert gas washout and spirometry versus structural lung disease in cystic fibrosis. Thorax. 2008 Feb;63(2):129-34. doi: 10.1136/thx.2007.077784. Epub 2007 Aug 3. PMID 17675316
- [Background] Owens CM, Aurora P, Stanojevic S, Bush A, Wade A, Oliver C, Calder A, Price J, Carr SB, Shankar A, Stocks J; London Cystic Fibrosis Collaboration. Lung Clearance Index and HRCT are complementary markers of lung abnormalities in young children with CF. Thorax. 2011 Jun;66(6):481-8. doi: 10.1136/thx.2010.150375. Epub 2011 Mar 21. PMID 21422040
- [Background] Hall GL, Logie KM, Parsons F, Schulzke SM, Nolan G, Murray C, Ranganathan S, Robinson P, Sly PD, Stick SM; AREST CF; Berry L, Garratt L, Massie J, Mott L, Poreddy S, Simpson S. Air trapping on chest CT is associated with worse ventilation distribution in infants with cystic fibrosis diagnosed following newborn screening. PLoS One. 2011;6(8):e23932. doi: 10.1371/journal.pone.0023932. Epub 2011 Aug 19. PMID 21886842
- [Background] Aurora P, Stanojevic S, Wade A, Oliver C, Kozlowska W, Lum S, Bush A, Price J, Carr SB, Shankar A, Stocks J; London Cystic Fibrosis Collaboration. Lung clearance index at 4 years predicts subsequent lung function in children with cystic fibrosis. Am J Respir Crit Care Med. 2011 Mar 15;183(6):752-8. doi: 10.1164/rccm.200911-1646OC. Epub 2010 Oct 8. PMID 20935113